CLINICAL TRIAL: NCT06132477
Title: Biometabolic Impact of Continuation of GLP-1 Agonists Following Bariatric
Brief Title: Impact GLP-1 Agonists Following Bariatric
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Society for Metabolic and Bariatric Surgery (Other)
Responsible Party: Principal Investigator, Andrew Wheeler, Assistant Professor of Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2098885
Record Dates: First submitted 2023-11-02; First posted 2023-11-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Morbid Obesity; Metabolic Syndrome; Diabetes Mellitus; Hypertension; Obstructive Sleep Apnea of Adult
Keywords: glp-1 agonist; Morbid Obesity; Bariatric Surgery; Metabolic syndrome; Diabetes Mellitus; Hypertension; Obstructive Sleep Apnea
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Diabetes Mellitus; Hypertension; Sleep Apnea, Obstructive | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Intervention Model Description: Patients will be continued on currently prescribed GLP-1 agonist after bariatric surgery or medication will be held
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 Agonist Group (Active Comparator): This cohort will consist of patients undergoing bariatric surgery who are currently receiving a GLP-1 Agonists for weight loss and/or diabetes management, that will be maintained on their preoperative dose of GLP-1 agonist following their bariatric surgery. This includes semaglutide, tirzepitide, among others. The dosage will be variable, but will be the same dose the patient is on prior to the bariatric surgery. Duration will be one of the aims of the study.
  Interventions: Drug: GLP-1 receptor agonist
- Non-GLP-1 Agonist Group (No Intervention): This cohort will consist of patients undergoing bariatric surgery who are currently receiving a GLP-1 Agonist for weight loss and/or diabetes management that will be required to stop taking their preoperative dose of GLP-1 agonist following their bariatric surgery. Dosage preoperative will be variable based on what the patient is currently taking, as well as the medication being taken.

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Randomized to continue or discontinue GLP-1 receptor agonists after bariatric surgery
  Other Names: GLP-1 agonists
  Arms: GLP-1 Agonist Group

SUMMARY:
Glucagon-like peptide 1 (GLP-1) is a hormone that helps regulate blood glucose levels through improved insulin sensitivity and release of insulin from the pancreas, control hunger, induce satiety and plays a role in the metabolic health of a person. GLP-1 receptor agonists (GLP1-RAs) have been shown to be effective in achieving weight loss in patients with type 2 diabetes while improving blood glucose control. Bariatric surgical procedures have been shown to be effective in treating obesity as well as superior to best medical therapy for treatment of diabetes not just through restriction of calories but also through a positive impact in modifications of gut hormones, changes in circulating bile acids, modifications in the gut microflora as well as other undefined mechanisms. The combined benefits of GLP1-RAs with bariatric surgery have only been studied to a limited effect. In this randomized trial, the effects of continuation or discontinuation of GLP1-RA therapy in patients undergoing bariatric surgery will be determined. We will compare changes in weight, metabolic determinants including circulating bile acids and gut microbiome, psychological determinants of eating behavior, and adverse side effects in patients who continue vs discontinue therapy. Given differences in metabolic and clinical outcomes in patients undergoing vertical sleeve gastrectomy (VSG) and Roux-en-Y gastric bypass (RYGB), both surgical groups will be examined. The study will be conducted at a high volume bariatric surgical program where patients will undergo randomization at the time of final clinic visit prior to surgery to continue or discontinue GLP1-RA. It is hypothesized that participants who continue GLP1-RA therapy after bariatric surgery will lose more weight with improved blood glucose control than those who discontinue therapy. Furthermore, changes in gut microbiome and circulating bile acids, known determinants of metabolic health, will be modified to a differential extent in those who are on GLP1-RAs vs those where GLP1-RAs are discontinued. Understanding the role these medications play in not only clinical outcomes after metabolic surgery but potential metabolic mechanisms by which surgery improves patient's metabolic health could help people with obesity and type 2 diabetes make informed decisions about their treatment options as well as advise providers on the continuation of these medications in the perioperative and postoperative period.

DETAILED DESCRIPTION:
Preliminary Work To date we have established a randomized controlled clinical trial where we are comparing groups of patients with variable lengths of biliopancreatic limb lengths during gastric bypass. VSG patients serve as a control surgical group, and we have gathered both serum and stool in over 200 patients. We have collaborated with both the institutional metagenomics and proteomics centers to process samples and evaluate bile acid synthesis and stool microbiome content. This trial has successful IRB approval for the project through the University of Missouri-Columbia IRB (#2058104) as well as registered the study with clinicaltrials.gov (NCT04841057).

Recruitment and Randomization:

1. Meet inclusion criteria and do not have any exclusion criteria
2. Meet all criteria per standard practice to qualify for surgery
3. Taking a GLP-1 agonist at time of consenting as part of their medical care apart from the research protocol
4. Recruitment will occur at the time of the preoperative education class which is the final visit prior to surgery. At this point patients will have determined whether or not they desire to have a sleeve gastrectomy or gastric bypass. For those who are taking a GLP-1 agonist they will be offered the ability to participate in the study.

Randomization of patients and surgical technique. A total of two groups will be utilized. Eligible patients will include those taking a GLP-1 agonist at the time of surgery. These patient will be randomized to either continuation of the GLP-1 agonist or discontinuation of the GLP-1 agonist. Surgical patients will include those undergoing sleeve gastrectomy, gastric bypass, duodenal switch, or revisional surgery.

Recruitment Site Weight Management and Metabolic Center Preoperative and post-operative weight loss surgery patients as well as non-surgical weight management patients are seen by providers at the Weight Management and Metabolic Center, a part of MU Health Care. Patients will undergo standard screening for medical and surgical history per any preoperative weight loss surgery patient. Per our standard protocol all patients will have a full set of nutrition labs which includes basic labs including complete blood count and complete metabolic profile as well as vitamin and nutrient labs.

Consent Process:

Each patient will be approached before the weight loss or bariatric surgery or during their care for medical weight loss or when being evaluated for non-weight loss surgery. In addition, Written Consent and HIPPA form consent will be provided for the patient to review, and one of the research staff listed on the local IRB will be available to answer any questions after the patient has sufficient time to review the consent.

Number of anticipated subjects:

Sample size for randomization to two groups will be 150 patients. This is based on power analysis to have an 80% power to detect a difference in percentage of excess body weight loss with a probability of a Type 1 error rate of 5%. This will provide adequate patients given several different procedures that will be performed on patients in each group and an attrition rate of 30% who do not follow through with either follow-up appointments or adherence to their randomization status/group.

Sample size was determined based on previously published literature. This is an appropriate number to demonstrate a statistical difference in weight loss, the primary end goal.

Study Procedures/ Design/ Treatment Plan:

Patients will be recruited for approximately 5 years to gather the appropriate sample size. Because each patient will have samples collected for 5 years, it will be approximately 10 years from last patient enrolled until study is completed.

Surgical Procedures Each patient will decide which surgical procedure he/she desires after the initial consultation with the surgeon.

A gastric bypass will be performed using our standard technique. In brief, all procedures will be performed laparoscopically as is standard practice. Specifically, at our institution, the gastric pouch will be constructed with a linear stapler approximately 5 cm long and 3 cm wide. The gastrojejunostomy anastomosis will be constructed either with a 25 mm circular stapler or a linear stapler. The linear stapler common gastroenterotomy will be closed in a running 2 layer manner to narrow to approximately 13-15 mm. The jejunojeunostomy will be created with a liner stapler after creation of BPL length of 100 cm and an alimentary limb length of 125 cm which will be connected to the gastric pouch via the gastrojejunostomy. The remaining small bowel, which will represent the common small bowel channel will also be measured. Measurements will be achieved in a standard manner.

Patients undergoing a sleeve gastrectomy will undergo a procedure to laparoscopically resect and remove approximately 80% by volume of the outer portion of the stomach. At our institution, specifically the sleeve gastrectomy is performed using a bougie as an intraluminal template for sizing purposes. The bougie is either 36 or 40 French per our usual practice.

Medication Use Protocol

1. Currently, continuation or discontinuation of GLP-1 agonists after bariatric surgery has not been established as standard of care and is at the discretion of the medical team (surgical or medical). No GLP-1 agonists will be initiated postoperatively if not taking one of these medications when having bariatric surgery.
2. All GLP-1 agonists will be stopped 1 weeks before bariatric surgery in line with current recommendations by the American Society of Anesthesiologists.
3. Following bariatric surgery to avoid missing a dose, the dose the patient is currently taken will be continued.
4. In the event the patient develops significant side effects that are intolerable by the patient and outline below, appropriate dose modification will occur
5. Only patients who are taking GLP-1 agonists as part of routine medical care will be included in the study. The current standard of care regarding continuation or cessation of GLP-1 agonists has not been established and is up to individual providers including primary care physicians or specialists prescribing these medications or the surgeon performing the bariatric procedure.

Preoperative and Postoperative Visits

* Routine care: all patients will have preoperative visits required to qualify for weight loss surgery. These visits are part of routine care. At one of the final visits prior to the procedure, routine laboratory studies will be performed. When the patient is able labs will be drawn at the time of routine laboratory studies. The additional labs will be paid for by the study and the routine studies billed to patient/insurance company
* Postoperative visits will be performed as per routine care at 1 week, 1 month, 3 months, 6 months and then annually thereafter. Data from these visits will be used for the research study
* Blood will be drawn at 3 month visit, 6 month visit and annual visits.

Specimen Collection

* Samples will be collected based on the below protocols. Samples including blood, stool, and solid tissue will be collected from all groups. Following collection, samples will be transferred to the laboratory using the labs well established protocol.
* These samples will be stored in the following manner:
* Following sample collection, the samples will be labelled with a deidentified label and sample code entered into a database. A separate database will be maintained by research staff
* Any other clinical data will be kept in a separate database with corresponding code to the pathologic specimen database. This clinical database will be maintained by research staff in the Department of Surgery. REDCap™ is a secure online web-based application that can be used to store clinical information to create a clinical database. REDCap will include a field that corresponds to the code entered into the tissue database maintained by research staff
* Blood collection: at a hospital clinical lab located at University Hospital or affiliated institutions
* For stool collection, the patient will be provided a collection kit to collect the sample. They will be instructed to collect a sample and mail it to the research lab using institution approved methodology.
* For liver specimen collection, electrocautery or ultrasonic dissector will be used to excise a small wedge of liver specimen during the patient's weight loss procedure or other operation.
* For omentum collection, this will be harvested with electrocautery or ultrasonic dissector during the patients' operation.
* For subcutaneous fat, this will be harvested with electrocautery during the patient's operation from a skin incision created for completion of the operation.
* For small bowel, it will be taken only during those operations where bowel is routinely removed and discarded, such as during the gastric bypass.
* Bile will be collected from gallbladder during cholecystectomy or small bowel during gastric bypass. Bile will only be removed from the gallbladder when the patient is undergoing a cholecystectomy. After removal of the gallbladder, 10 cc of bile will be collected for research purposes.
* For stomach removed during sleeve gastrectomy this is removed at the time of the operation. A portion of the stomach will be removed for research specimen and the rest sent as a surgical specimen to the pathology laboratory

Clinical Data Collection

* A prospective clinical database will be maintained with relevant clinical data.
* In order to have relevant clinical data to allow for identification of the specimen and if relevant for planned research the research staff as mentioned above research staff listed on IRB will collect a limited amount of clinical data including name, date of birth, medical record number and procedure performed or medical weight loss as relevant.
* Any additional clinical data will be maintained by research staff within the Department of Surgery using RedCap TM or a spreadsheet located on a HIPAA compliant University of Missouri approved, cloud-based platform.
* The clinical database and specimen codes will be maintained research staff of the Department of Surgery at the University of Missouri School of Medicine where it will be maintained in a secure manner to protect identifiable patient data.
* This database will be deidentified for all HIPAA protected personal health information. This HIPAA protected health information will be kept in a separate database in a separate location that is password protected. It will also be maintained in a cloud-based platform. The two databases will be linked by a code with corresponding code linking the samples kept secure in a cloud-based platform and maintained by research staff
* Only research staff listed on IRB will have access to the key that allows identification of protected health information in the database
* Patients will be unblinded to which group they are in with regards to continuation or discontinuation of a GLP-1 agonist. Surgeons performing the operation will also be unblinded.

All patients will be performed for patients per routine care provided through metabolic and bariatric clinic. Regarding GLP-1 agonist therapy there is currently no standard of care whether to continue or discontinue their use after bariatric surgery.

Data Safety Monitoring Plan

The following additional variables will be included in the prospective database at the following follow-up visits (3 month, 6 months, 12 month, 24 months, 36 months, 48 months, and 60 months follow-up) and used to monitor for complications or adverse events:

1. Diagnosed protein calorie malnutrition
2. Presence of adverse GI side effects
3. Presence of excessive weight loss defined as BMI less than 20
4. Vitamin or micronutrient deficiencies

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years of age
2. Participation in care by one of the surgeons at MU Health Care
3. Undergoing surgical weight loss through the Weight Management and Metabolic Center
4. Body mass index of 30-80 kg/m2
5. Meet insurance criteria, as set forth by the patient's insurance policy, to qualify for coverage for weight loss surgery or as a self-pay patient for the weight loss procedure
6. Planned laparoscopic Roux-en-Y gastric bypass, sleeve gastrectomy, revisional weight loss surgery, or duodenal switch or modification of. If patients are not willing to be randomized they will not be enrolled as randomized but can still participate having samples collected.
7. Willingness to have blood collected before and after surgical procedure at defined points or at minimum have clinical data collected.
8. Willingness to have clinical data entered into a prospective database
9. Additional specimens collected as stated in the protocol will be offered but collection not mandated.

5. Taking a GLP-1 agonist as part of their routine medical care apart from any planned surgical procedure. The current standard of care regarding continuation or discontinuation of GLP-1 agonists has not been established and is at the discretion of members of the patient's medical team but to be included the patient and medical care team must be willing to continue or discontinue the GLP-1 agonist after surgery depending on the randomized group.

Exclusion Criteria:

1. Pregnant patient
2. Desire to not participate
3. Age less than 18
4. Patient fails to fulfill insurance mandated criteria and is not interested in paying cash for their procedure
5. Not taking a GLP-1 agonist as part of standard medical care
6. Unwilling to follow-up at required postoperative visits
7. Unwilling to stop GLP-1 agonist if randomized into group to stop GLP-1 agonist or unwilling to continue the GLP-1 agonist if randomized into that respective group. If chooses to continue or discontinue the medication apart from randomization the patient can still participate as a non-randomized participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Effect of GLP1-RA on weight loss | 6 months
  To investigate the effects of GLP1-RAs on weight loss reflected as change in BMI (kg per meter sq) in patients undergoing metabolic surgery
Effect of GLP1-RA on circulating bile acids and metabolites | 6 months
  Determine the impact of GLP1-RA on circulating bile acids and other metabolites
Effector of GLP1-RA on gut microbiome diversity | 6 months
  To determine the impact of GLP1-RAs after bariatric surgery on changes in the gut microbiome
Effect of GLP1-RA on satiety and hunger | 6 months
  To assess the impact of GLP-1 agonists on satiety and hunger in patients who undergo metabolic surgery. Scale will be a validated scoring system, "Daily Eats Questionnaire," with scores ranging from 0-10, with a 0 indicating no hunger, and 10 indicating extreme hunger
Effect of GLP1-RA on Glycemic control | 6 months
  HGBA1C levels will be measured at 3 and 6 months after surgery to determine if HGBA1C drops more in patients maintained on GLP1-RA

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wheeler, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will be collecting data on the participants in the study including glycemic control and weight loss. We will also including information on specimens which include bile acids, and microbiome. While at this time we do not have any plans to make individual participant data (IPD) available to other researchers, we are undecided.

REFERENCES:
- [Background] Lee SJ, Shin SW. Mechanisms, Pathophysiology, and Management of Obesity. N Engl J Med. 2017 Apr 13;376(15):1491-2. doi: 10.1056/NEJMc1701944. No abstract available. PMID 28406283
- [Background] Mouton AJ, Li X, Hall ME, Hall JE. Obesity, Hypertension, and Cardiac Dysfunction: Novel Roles of Immunometabolism in Macrophage Activation and Inflammation. Circ Res. 2020 Mar 13;126(6):789-806. doi: 10.1161/CIRCRESAHA.119.312321. Epub 2020 Mar 12. PMID 32163341
- [Background] Zhang Y, Liu J, Yao J, Ji G, Qian L, Wang J, Zhang G, Tian J, Nie Y, Zhang YE, Gold MS, Liu Y. Obesity: pathophysiology and intervention. Nutrients. 2014 Nov 18;6(11):5153-83. doi: 10.3390/nu6115153. PMID 25412152
- [Background] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Brethauer SA, Navaneethan SD, Aminian A, Pothier CE, Kim ES, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric surgery versus intensive medical therapy for diabetes--3-year outcomes. N Engl J Med. 2014 May 22;370(21):2002-13. doi: 10.1056/NEJMoa1401329. Epub 2014 Mar 31. PMID 24679060
- [Background] Blond E, Disse E, Cuerq C, Drai J, Valette PJ, Laville M, Thivolet C, Simon C, Caussy C. EASL-EASD-EASO clinical practice guidelines for the management of non-alcoholic fatty liver disease in severely obese people: do they lead to over-referral? Diabetologia. 2017 Jul;60(7):1218-1222. doi: 10.1007/s00125-017-4264-9. Epub 2017 Mar 28. PMID 28352941
- [Background] de Witte D, Wijngaarden LH, van Houten VAA, van den Dorpel MA, Bruning TA, van der Harst E, Klaassen RA, Niezen RA. Improvement of Cardiac Function After Roux-en-Y Gastric Bypass in Morbidly Obese Patients Without Cardiac History Measured by Cardiac MRI. Obes Surg. 2020 Jul;30(7):2475-2481. doi: 10.1007/s11695-020-04543-y. PMID 32198618
- [Background] Schauer DP, Feigelson HS, Koebnick C, Caan B, Weinmann S, Leonard AC, Powers JD, Yenumula PR, Arterburn DE. Bariatric Surgery and the Risk of Cancer in a Large Multisite Cohort. Ann Surg. 2019 Jan;269(1):95-101. doi: 10.1097/SLA.0000000000002525. PMID 28938270
- [Background] Pucci A, Batterham RL. Mechanisms underlying the weight loss effects of RYGB and SG: similar, yet different. J Endocrinol Invest. 2019 Feb;42(2):117-128. doi: 10.1007/s40618-018-0892-2. Epub 2018 May 5. PMID 29730732
- [Background] Sakran N, Soifer K, Hod K, Sherf-Dagan S, Soued S, Kessler Y, Adelson D, Biton R, Buchwald JN, Goitein D, Raziel A. Long-term Reported Outcomes Following Primary Laparoscopic Sleeve Gastrectomy. Obes Surg. 2023 Jan;33(1):117-128. doi: 10.1007/s11695-022-06365-6. Epub 2022 Nov 28. PMID 36441488
- [Background] Cooper TC, Simmons EB, Webb K, Burns JL, Kushner RF. Trends in Weight Regain Following Roux-en-Y Gastric Bypass (RYGB) Bariatric Surgery. Obes Surg. 2015 Aug;25(8):1474-81. doi: 10.1007/s11695-014-1560-z. PMID 25595383
- [Background] Abel SA, English WJ, Duke MC, Williams DB, Aher CV, Broucek JR, Spann MD. Benefits of Adjuvant Medical Weight Loss Intervention in Setting of Weight Regain and Inadequate Weight Loss After Weight Loss Surgery. Am Surg. 2023 May;89(5):1857-1863. doi: 10.1177/00031348221078957. Epub 2022 Mar 22. PMID 35317659
- [Background] Blundell J, Finlayson G, Axelsen M, Flint A, Gibbons C, Kvist T, Hjerpsted JB. Effects of once-weekly semaglutide on appetite, energy intake, control of eating, food preference and body weight in subjects with obesity. Diabetes Obes Metab. 2017 Sep;19(9):1242-1251. doi: 10.1111/dom.12932. Epub 2017 May 5. PMID 28266779
- [Background] Astrup A, Carraro R, Finer N, Harper A, Kunesova M, Lean ME, Niskanen L, Rasmussen MF, Rissanen A, Rossner S, Savolainen MJ, Van Gaal L; NN8022-1807 Investigators. Safety, tolerability and sustained weight loss over 2 years with the once-daily human GLP-1 analog, liraglutide. Int J Obes (Lond). 2012 Jun;36(6):843-54. doi: 10.1038/ijo.2011.158. Epub 2011 Aug 16. PMID 21844879
- [Background] Hindso M, Hedback N, Svane MS, Moller A, Martinussen C, Jorgensen NB, Dirksen C, Gasbjerg LS, Kristiansen VB, Hartmann B, Rosenkilde MM, Holst JJ, Madsbad S, Bojsen-Moller KN. The Importance of Endogenously Secreted GLP-1 and GIP for Postprandial Glucose Tolerance and beta-Cell Function After Roux-en-Y Gastric Bypass and Sleeve Gastrectomy Surgery. Diabetes. 2023 Mar 1;72(3):336-347. doi: 10.2337/db22-0568. PMID 36478039
- [Background] Garvey WT, Mechanick JI, Brett EM, Garber AJ, Hurley DL, Jastreboff AM, Nadolsky K, Pessah-Pollack R, Plodkowski R; Reviewers of the AACE/ACE Obesity Clinical Practice Guidelines. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY COMPREHENSIVE CLINICAL PRACTICE GUIDELINES FOR MEDICAL CARE OF PATIENTS WITH OBESITY. Endocr Pract. 2016 Jul;22 Suppl 3:1-203. doi: 10.4158/EP161365.GL. Epub 2016 May 24. PMID 27219496
- [Background] Wirunsawanya K, Chittimoju S, Fantasia KL, Modzelewski KL, Steenkamp D, Alexanian SM. Insulin Requirements in Patients With Type 2 Diabetes Undergoing Bariatric Surgery in the Inpatient Setting and Upon Discharge: A Single-Center Retrospective Analysis of Insulin Management Strategies. Endocr Pract. 2021 Jun;27(6):538-544. doi: 10.1016/j.eprac.2020.12.014. Epub 2021 Jan 11. PMID 34016530
- [Background] Sarma S, Palcu P. Weight loss between glucagon-like peptide-1 receptor agonists and bariatric surgery in adults with obesity: A systematic review and meta-analysis. Obesity (Silver Spring). 2022 Nov;30(11):2111-2121. doi: 10.1002/oby.23563. PMID 36321278
- [Background] Jensen AB, Renstrom F, Aczel S, Folie P, Biraima-Steinemann M, Beuschlein F, Bilz S. Efficacy of the Glucagon-Like Peptide-1 Receptor Agonists Liraglutide and Semaglutide for the Treatment of Weight Regain After Bariatric surgery: a Retrospective Observational Study. Obes Surg. 2023 Apr;33(4):1017-1025. doi: 10.1007/s11695-023-06484-8. Epub 2023 Feb 11. PMID 36765019
- [Background] Llewellyn DC, Logan Ellis H, Aylwin SJB, Ostarijas E, Green S, Sheridan W, Chew NWS, le Roux CW, Miras AD, Patel AG, Vincent RP, Dimitriadis GK. The efficacy of GLP-1RAs for the management of postprandial hypoglycemia following bariatric surgery: a systematic review. Obesity (Silver Spring). 2023 Jan;31(1):20-30. doi: 10.1002/oby.23600. Epub 2022 Dec 10. PMID 36502288
- [Background] Guarino D, Moriconi D, Mari A, Rebelos E, Colligiani D, Baldi S, Anselmino M, Ferrannini E, Nannipieri M. Postprandial hypoglycaemia after Roux-en-Y gastric bypass in individuals with type 2 diabetes. Diabetologia. 2019 Jan;62(1):178-186. doi: 10.1007/s00125-018-4737-5. Epub 2018 Oct 12. PMID 30315341
- [Background] Madsbad S. Review of head-to-head comparisons of glucagon-like peptide-1 receptor agonists. Diabetes Obes Metab. 2016 Apr;18(4):317-32. doi: 10.1111/dom.12596. Epub 2015 Dec 29. PMID 26511102
- [Background] Hurtado A MD, Acosta A. Precision Medicine and Obesity. Gastroenterol Clin North Am. 2021 Mar;50(1):127-139. doi: 10.1016/j.gtc.2020.10.005. Epub 2021 Jan 5. PMID 33518159
- [Background] de Vos WM, Tilg H, Van Hul M, Cani PD. Gut microbiome and health: mechanistic insights. Gut. 2022 May;71(5):1020-1032. doi: 10.1136/gutjnl-2021-326789. Epub 2022 Feb 1. PMID 35105664
- [Background] Shapiro H, Kolodziejczyk AA, Halstuch D, Elinav E. Bile acids in glucose metabolism in health and disease. J Exp Med. 2018 Feb 5;215(2):383-396. doi: 10.1084/jem.20171965. Epub 2018 Jan 16. PMID 29339445
- [Background] Jonsson I, Bojsen-Moller KN, Kristiansen VB, Veedfald S, Wewer Albrechtsen NJ, Clausen TR, Kuhre RE, Rehfeld JF, Holst JJ, Madsbad S, Svane MS. Effects of Manipulating Circulating Bile Acid Concentrations on Postprandial GLP-1 Secretion and Glucose Metabolism After Roux-en-Y Gastric Bypass. Front Endocrinol (Lausanne). 2021 May 14;12:681116. doi: 10.3389/fendo.2021.681116. eCollection 2021. PMID 34084153
- [Background] Pournaras DJ, Glicksman C, Vincent RP, Kuganolipava S, Alaghband-Zadeh J, Mahon D, Bekker JH, Ghatei MA, Bloom SR, Walters JR, Welbourn R, le Roux CW. The role of bile after Roux-en-Y gastric bypass in promoting weight loss and improving glycaemic control. Endocrinology. 2012 Aug;153(8):3613-9. doi: 10.1210/en.2011-2145. Epub 2012 Jun 6. PMID 22673227
- [Background] Chaudhari SN, Luo JN, Harris DA, Aliakbarian H, Yao L, Paik D, Subramaniam R, Adhikari AA, Vernon AH, Kilic A, Weiss ST, Huh JR, Sheu EG, Devlin AS. A microbial metabolite remodels the gut-liver axis following bariatric surgery. Cell Host Microbe. 2021 Mar 10;29(3):408-424.e7. doi: 10.1016/j.chom.2020.12.004. Epub 2021 Jan 11. PMID 33434516
- [Background] Jendle J, Hyotylainen T, Oresic M, Nystrom T. Pharmacometabolomic profiles in type 2 diabetic subjects treated with liraglutide or glimepiride. Cardiovasc Diabetol. 2021 Dec 17;20(1):237. doi: 10.1186/s12933-021-01431-2. PMID 34920733
- [Background] Madsen MSA, Holm JB, Palleja A, Wismann P, Fabricius K, Rigbolt K, Mikkelsen M, Sommer M, Jelsing J, Nielsen HB, Vrang N, Hansen HH. Metabolic and gut microbiome changes following GLP-1 or dual GLP-1/GLP-2 receptor agonist treatment in diet-induced obese mice. Sci Rep. 2019 Oct 30;9(1):15582. doi: 10.1038/s41598-019-52103-x. PMID 31666597
- [Background] Ocana-Wilhelmi L, Martin-Nunez GM, Ruiz-Limon P, Alcaide J, Garcia-Fuentes E, Gutierrez-Repiso C, Tinahones FJ, Moreno-Indias I. Gut Microbiota Metabolism of Bile Acids Could Contribute to the Bariatric Surgery Improvements in Extreme Obesity. Metabolites. 2021 Oct 27;11(11):733. doi: 10.3390/metabo11110733. PMID 34822391
- [Background] Gentile JKA, Oliveira KD, Pereira JG, Tanaka DY, Guidini GN, Cadona MZ, Siriani-Ribeiro DW, Perondini MT. THE INTESTINAL MICROBIOME IN PATIENTS UNDERGOING BARIATRIC SURGERY: A SYSTEMATIC REVIEW. Arq Bras Cir Dig. 2022 Dec 19;35:e1707. doi: 10.1590/0102-672020220002e1707. eCollection 2022. PMID 36542005
- [Background] Thakur U, Bhansali A, Gupta R, Rastogi A. Liraglutide Augments Weight Loss After Laparoscopic Sleeve Gastrectomy: a Randomised, Double-Blind, Placebo-Control Study. Obes Surg. 2021 Jan;31(1):84-92. doi: 10.1007/s11695-020-04850-4. Epub 2020 Jul 12. PMID 32656729
- [Background] Chaar ME, Lundberg P, Stoltzfus J. Thirty-day outcomes of sleeve gastrectomy versus Roux-en-Y gastric bypass: first report based on Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program database. Surg Obes Relat Dis. 2018 May;14(5):545-551. doi: 10.1016/j.soard.2018.01.011. Epub 2018 Jan 13. PMID 29551470
- [Background] Lewis CA, de Jersey S, Seymour M, Hopkins G, Hickman I, Osland E. Iron, Vitamin B12, Folate and Copper Deficiency After Bariatric Surgery and the Impact on Anaemia: a Systematic Review. Obes Surg. 2020 Nov;30(11):4542-4591. doi: 10.1007/s11695-020-04872-y. Epub 2020 Aug 12. PMID 32785814
- [Background] James H, Lorentz P, Collazo-Clavell ML. Patient-Reported Adherence to Empiric Vitamin/Mineral Supplementation and Related Nutrient Deficiencies After Roux-en-Y Gastric Bypass. Obes Surg. 2016 Nov;26(11):2661-2666. doi: 10.1007/s11695-016-2155-7. PMID 27038046
- [Background] Meyer Mikalsen S, Aaseth J, Flaten TP, Whist JE, Bjorke-Monsen AL. Essential trace elements in Norwegian obese patients before and 12 months after Roux-en-Y gastric bypass surgery: Copper, manganese, selenium and zinc. J Trace Elem Med Biol. 2020 Dec;62:126650. doi: 10.1016/j.jtemb.2020.126650. Epub 2020 Sep 21. PMID 33011630
- [Background] Arias PM, Domeniconi EA, Garcia M, Esquivel CM, Martinez Lascano F, Foscarini JM. Micronutrient Deficiencies After Roux-en-Y Gastric Bypass: Long-Term Results. Obes Surg. 2020 Jan;30(1):169-173. doi: 10.1007/s11695-019-04167-x. PMID 31502183
- See also: Body Mass Index as a Patient Selection Criterion for Kidney Transplant — https://doi.org/10.15367/ch.v1i1.302